CLINICAL TRIAL: NCT04940533
Title: Pharmacokinetics of CFTR Modulators in Pregnant Individuals and in Postpartum Breastfeeding Mothers
Status: Not yet recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PACCS-2020-28860-1
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis; Pregnancy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving CFTR modulator therapy - Trikafta: This is a single arm study. Participants in this study are receiving CFTR modulator therapy.

SUMMARY:
This study aims to evaluate the pharmacokinetic changes during pregnancy, postpartum, and in breast milk in cystic fibrosis patients receiving a cystic fibrosis transmembrane conductance regulator (CTFR) modulator, including Elexacaftor, Tezacaftor, Ivacaftor, or Lumacaftor.

DETAILED DESCRIPTION:
The advent of cystic fibrosis transmembrane conductance regulator (CFTR) therapy has significantly increased the life expectancy for individuals with cystic fibrosis (CF).

As a result, adults with CF are more likely to have families than they have in the past.

Although the overall pregnancy rate among women with CF age 18-44 is declining (mirroring trends in the general population), the overall number of pregnancies is increasing due to the increasing number of adults with CF. However, little is known about CFTR modulator use in pregnant or breastfeeding mothers, as outlined in a recent review of CF-therapies in pregnant and breastfeeding women. Presently, there is one report of an uncomplicated pregnancy during ivacaftor use, and one case of a successful pregnancy in a woman who was maintained on lumacaftor/ivacaftor with reported maternal and fetal drug levels. In this study, we aim to study the pharmacokinetics of CFTR modulators in pregnancy as well as while breastfeeding.

This information will hopefully improve counseling while offering them for CF patients given the tremendous improvements seen in non-pregnant adults.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age and older
* Female who has a diagnosis of cystic fibrosis
* Female who is taking cystic fibrosis transmembrane conductance regulator (CFTR) modulator medication during pregnancy and postpartum

Exclusion Criteria:

* Female < 18 years of age
* Female with cystic fibrosis who is not taking cystic fibrosis transmembrane conductance regulator (CFTR) modulator medication during pregnancy and postpartum
* Participant has contraindication to breastfeeding or not planning to breastfeed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females receiving cystic fibrosis transmembrane conductance regulator (CFTR) modulation therapy who are pregnant or breastfeeding.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in levels of CTFR modulator in blood | approximately 9 months
  Quantification of CTFR modulator in blood will be performed using Liquid Chromatography-Mass Spectrometry (LC-MS) and reported in units of ng/kg. Blood will be collected every 3 months during pregnancy and at the sampling of breast milk 0-4 days after giving birth.
Change in levels of CTFR modulator in breast milk | 4 days
  Quantification of CTFR modulator in blood will be performed using Liquid Chromatography-Mass Spectrometry (LC-MS) and reported in units of ng/ml. Breast milk will be collected following feeding of the infant 0-4 days following birth of the infant.
Change in levels of CTFR modulator in umbilical cord blood | at birth of the infant
  Quantification of CTFR modulator in blood will be performed using Liquid Chromatography-Mass Spectrometry (LC-MS) and reported in units of ng/kg. Umbilical cord blood will be collected once at the time the infant is born.

CONTACTS AND LOCATIONS:
Overall Officials: Jagadish Patil, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No